CLINICAL TRIAL: NCT02734303
Title: Study to Estimate Radiation Doses and Cancer Risks From Radioactive Fallout From the Trinity Nuclear Test
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916083; 16-C-N083
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Cancers
Keywords: Dietary Radioactivity; Dietary Assessment; Retrospective Recall; Focus Group
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Potentially Exposed NM Residents: residents of the state of New Mexico (NM) potentially exposed to radioactive fallout fromthe Trinity nuclear test conducted in 1945

SUMMARY:
Background:

The first nuclear bomb test took place in New Mexico in July 1945. This was called the Trinity test. Researchers want to learn how it affected the health of people who lived in New Mexico at the time of the test. To do this, they want to learn about the diet and daily life of those people at that time. They want to study Native Americans, Hispanic/Latinos, and non-Hispanic/Latino whites.

Objective:

To learn about the health risks for people who may have been exposed to radiation from the Trinity nuclear test.

Eligibility:

People who:

* Are Native American, Hispanic/Latino, or non-Hispanic white
* Are age 70 and older
* Lived near the fallout region of the Trinity test and know about lifestyle and dietary patterns in New Mexico in the 1940s and 1950s

Design:

Participants will be screened with a questionnaire.

Participants will answer questions in an interview or a focus group. This will be at a place like an office, tribal or community center, or library. It will take up to 2 hours. The interview or group session will include:

* Questions about their and their family members activities and eating habits in the 1940s and 1950s
* A card-sorting exercise: There will be cards with pictures and names of certain foods. They will sort the cards into 2 piles: those that were consumed and those that were not.
* Filling out a chart of their family members and the foods they ate

If participants give permission, their interview or group session will be recorded.

...

DETAILED DESCRIPTION:
Over the last four decades, assessments of health risks based on estimated radiation doses received by the public have been completed for all major U.S. nuclear testing sites and nuclear fuel cycle facilities in the U.S. except for the Trinity test. This research plan is for a radiationrelated cancer risk projection study for the residents of the state of New Mexico (NM) potentially exposed to radioactive fallout from the Trinity nuclear test conducted in 1945. Data to be collected on diet and lifestyle from the three main ethnic groups in NM (white, Hispanic, and Native American) via focus groups and key informant interviews will be used to derive means and ranges of exposure-related parameters for a dose assessment and risk projection. As preliminary work to this proposal, in 2014 we conducted a pilot study to obtain information from 9 key informants (maximum number allowed under OMB regulations prior to clearance) determined that the elders could recall the relevant time period and relevant lifestyle practices. This work established that it is possible to: 1) locate elderly representative of the ethnic groups, 2) assemble groups of members of tribal, a n d Hispanic/Latino communities in New Mexico who were alive in 1945 at the time of the test to participate in focus groups, and 3) obtain lifestyle and diet information to be used for refining focus group interviewing tools. Due to the successful completion of the pilot phase, here we are proposing a second phase to collect data, on a larger scale, via focus group and individual interviews, on lifestyle and diet from up to 150 Native American, Hispanic/Latino, and non-Hispanic white participants living in New Mexico who were alive at the time of the Trinity detonation (currently greater than or equal to 70 years old). The data collected in the proposed study will allows us to estimate exposure-related parameter values that can be used in fallout dose assessment models to estimate external and internal radiation doses to representative persons in all counties in New Mexico by ethnicity, gender, and age. Those doses will be used with published risk models and coupled with literature-derived parameters on risk/unit dose to project the excess cancers (per 1,000 persons within each strata) expected. Endpoints are leukemia, thyroid cancer, stomach cancer, and colon cancer.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Hispanic/Latino, non-Hispanic White or Native American
* 70 years or older (Alive in 1945)
* Resided in New Mexico or on one of New Mexico s tribal reservations (if Native American) during the 1940s and 1950s
* Ideally, helped to care for children in his or her community during the 1940s
* Potential focus group members an d key informants may include any of the following:

  * Community elders, tribal members, and people with first hand knowledge of food practices in New Mexico in the 1940s or 1950s.
  * Individuals must self-identify as a New Mexico tribal community member, Hispanic/Latino or non-Hispanic white in order to participate

in an interview, and have firsthand knowledge about lifestyle and dietary patterns in New Mexico during the 1940s or 1950s.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Residents of the state of New Mexico (NM) potentially exposed to radioactive fallout from the Trinity nuclear test conducted in 1945.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
risk assessment | Cumulative since 1945 exposure
  prediction of number of excess cancers of: colon, lung, active bone marrow, stomach, and thyroid

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Simon, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Simon SL, Bouville A. Radiation doses to local populations near nuclear weapons test sites worldwide. Health Phys. 2002 May;82(5):706-25. doi: 10.1097/00004032-200205000-00016. PMID 12003020
- [Background] Schwerin M, Schonfeld S, Drozdovitch V, Akimzhanov K, Aldyngurov D, Bouville A, Land C, Luckyanov N, Mabuchi K, Semenova Y, Simon S, Tokaeva A, Zhumadilov Z, Potischman N. The utility of focus group interviews to capture dietary consumption data in the distant past: dairy consumption in Kazakhstan villages 50 years ago. J Dev Orig Health Dis. 2010 Jun;1(3):192-202. doi: 10.1017/S2040174410000243. PMID 24286002